CLINICAL TRIAL: NCT02182635
Title: A Phase III Long-term Study of Ba253BINEB in Patients With COPD
Brief Title: Ba253BINEB in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54.561
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (1):
- Ba253BINEB (Experimental)
  Interventions: Drug: Ba253BINEB

INTERVENTIONS:
Drug: Ba253BINEB

SUMMARY:
The objective of this study is to investigate the long-term safety of Ba253BINEB. Secondarily the long-term efficacy of Ba253BINEB is also investigated.

ELIGIBILITY:
Inclusion Criteria:

The patients with COPD (chronic bronchitis, emphysema) and who satisfy the following criteria

1. Patients with FEV1.0/FVC (Forced vital capacity) of <= 70% in the screening test and whose symptoms are stable
2. Patients aged >= 40 years or older
3. Patients must be able to understand the patient information form

Exclusion Criteria:

1. Patients complicated with bronchial asthma, making the assessment of drug efficacy against COPD difficult
2. Patients who have taken an long acting corticosteroids(i.m.) within 1 month before the study
3. Patients using oral corticosteroid medication at a dose in excess of the equivalent 5 mg/day of prednisolone
4. Patients with glaucoma
5. Patients who have prostatic hypertrophy
6. Patients with hypersensitivity to anticholinergic drugs
7. Patients with serious hepatic disease, kidney disease or heart disorder and who are judged by the investigator as inappropriate as the subjects of study
8. Women who are pregnant or who may become pregnant, or nursing women
9. Patients who are judged by the investigator as inappropriate as the subjects of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 1998-08; Primary Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events | Up to 28 weeks
Number of patients with significant changes from baseline in vital signs (blood pressure, heart rate) | Baseline, up to week 28
Number of patients with abnormal changes from baseline in electrocardiogram (ECG) | Baseline, up to week 28
Number of patients wiht abnormal changes from baseline in laboratory tests | Baseline, up to week 28

SECONDARY OUTCOMES:
Change from baseline in FEV1 (Forced expiratory volume in one second) | Baseline, up to week 28
Change from baseline in COPD symptom scoring (cough, sputum amount, shortness of breath, nocturnal sleep) | Baseline, up to week 28
Physician's global evaluation (overall improvement) | Up to week 28
Patient's impression | Week 28
Physician's global evaluation (final improvement) | Week 28